CLINICAL TRIAL: NCT00083239
Title: Study of Talabostat in Advanced Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Point Therapeutics (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTH-301
Record Dates: First submitted 2004-05-14; First posted 2004-05-18 (Estimated); Last update posted 2007-06-08 (Estimated); Status verified 2007-06

CONDITIONS: Melanoma; Skin Cancer
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — talabostat; Tablets

INTERVENTIONS:
Drug: talabostat (PT-100) tablets

SUMMARY:
The purpose of this study is to assess the antitumor activity and safety of talabostat in patients with metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed melanoma that is metastatic (unresectable Stage IV per AJCC 2002)
* Patients with measurable disease defined as at least one measurable index lesion with clearly defined margins
* ECOG Performance Status of 0, 1, or 2
* Expected survival ≥12 weeks
* Written informed consent

Exclusion Criteria:

* More than 1 prior chemotherapy or biotherapy regimen for Stage IV melanoma
* Radiation therapy to >50% of the bone marrow. Patients must not have had prior radiotherapy to index lesions unless they have clearly progressive disease in this site or there is measurable disease outside the area of prior radiation.
* Clinically significant laboratory abnormalities
* CNS metastases
* Any malignancy within the 5 years immediately prior to the first dose of study medication with the exception of basal cell or non-metastatic squamous cell carcinoma of the skin, and carcinoma in-situ of the cervix
* The need for chronic (i.e., >7 days) oral or intravenous corticosteroid therapy
* Any comorbidity or condition which, in the opinion of the investigator, may interfere with the assessments and procedures of this protocol
* Patients who are within 30 days of chemotherapy, radiation therapy, immunotherapy, or other investigational medication for melanoma. Patients must have recovered from all of the side effects of treatment in order to be enrolled.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Mary Crowley Medical Research Center, Dallas, Texas